CLINICAL TRIAL: NCT05495438
Title: Impact and Safety of AI in Decision Making in the ICU: a Simulation Experiment
Acronym: ICU
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University of York (Other)
Responsible Party: Sponsor
Other Study IDs: 22CX7592
Record Dates: First submitted 2022-08-04; First posted 2022-08-10 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Sepsis
Keywords: Artificial Intelligence
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU Clinicians
  Interventions: Other: Hypothetical AI

INTERVENTIONS:
Other: Hypothetical AI — n/a - There is no intervention. Clinicians will review the suggestions of a hypothetical AI

SUMMARY:
The impact of deploying artificial intelligence (AI) in healthcare settings in unclear, in particular with regards to how it will influence human decision makers. Previous research demonstrated that AI alerts were frequently ignored (Kamal et al., 2020 ) or could lead to unexpected behaviour with worsening of patient outcomes (Wilson et al., 2021 ). On the other hand, excessive confidence and trust placed in the AI could have several adverse consequences including ability to detect harmful AI decisions, leading to patient harm as well as human deskilling. Some of these aspects relate to automation bias.

In this simulation study, the investigators intend to measure whether medical decisions in areas of high clinical uncertainty are modified by the use of an AI-based clinical decision support tool. How the dose of intravenous fluids (IVF) and vasopressors administered by doctors in adult patients with sepsis (severe infection with organ failure) in the ICU), changes as a result of disclosing the doses suggested by a hypothetical AI will be measured. The area of sepsis resuscitation is poorly codified, with high uncertainty leading to high variability in practice. This study will not specifically mention the AI Clinician (Komorowski et al., 2018). Instead, the investigators will describe a hypothetical AI for which there is some evidence of effectiveness on retrospective data in another clinical setting (e.g. a model that was retrospectively validated using data from a different country than the source data used for model training) but no prospective evidence of effectiveness or safety. As such, it is possible for this hypothetical AI to provide unsafe suggestions. The investigators will intentionally introduce unsafe AI suggestions (in random order), to measure the sensitivity of our participants at detecting these.

DETAILED DESCRIPTION:
The impact of deploying artificial intelligence (AI) in healthcare settings in unclear, in particular with regards to how it will influence human decision makers. Previous research demonstrated that AI alerts were frequently ignored (Kamal et al., 2020 ) or could lead to unexpected behaviour with worsening of patient outcomes (Wilson et al., 2021 ). On the other hand, excessive confidence and trust placed in the AI could have several adverse consequences including ability to detect harmful AI decisions, leading to patient harm as well as human deskilling. Some of these aspects relate to automation bias.

In this simulation study, the investigators intend to measure whether medical decisions in areas of high clinical uncertainty are modified by the use of an AI-based clinical decision support tool. How the dose of intravenous fluids (IVF) and vasopressors administered by doctors in adult patients with sepsis (severe infection with organ failure) in the ICU), changes as a result of disclosing the doses suggested by a hypothetical AI will be measured. The area of sepsis resuscitation is poorly codified, with high uncertainty leading to high variability in practice. This study will not specifically mention the AI Clinician (Komorowski et al., 2018). Instead, the investigators will describe a hypothetical AI for which there is some evidence of effectiveness on retrospective data in another clinical setting (e.g. a model that was retrospectively validated using data from a different country than the source data used for model training) but no prospective evidence of effectiveness or safety. As such, it is possible for this hypothetical AI to provide unsafe suggestions. The investigators will intentionally introduce unsafe AI suggestions (in random order), to measure the sensitivity of our participants at detecting these.

The investigators will examine what participant characteristics are linked with an increase likelihood of being influenced by the AI, and conduct a number of pre-specified subgroup analyses, e.g. junior versus senior ICU doctors, and separating those with a positive or a negative attitude towards AI.

ELIGIBILITY:
Inclusion Criteria:

* Junior (senior house officer) or senior (registrar/fellow/consultant) ICU doctor

Exclusion Criteria:

* Participants not meeting the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Junior (senior house officer) or senior (registrar/fellow/consultant) ICU doctor
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Influence of AI on ICU Clinicians | 3 months
  Influence of AI on ICU Clinicians, this will be divided into the following categories: overall and stratified by safe/unsafe, junior/senior and positive/negative attitude towards AI.

SECONDARY OUTCOMES:
Participants' characteristics | 3 months
  What are the characteristics of those taking part in the simulation and how does this affect decision making.
Trust in AI | 3 months
  How much do ICU clinicians trust the AI system.
Confidence in participants' decisions | 3 months
  How much confidence do clinicians place in the AI system
Proportion of time with attention on AI explanation | 3 months
  Where is attention focused during the simulation

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Komorowski, MD, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Hospitals NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be reviewed by the study team.